CLINICAL TRIAL: NCT06597084
Title: Prevention of Epilepsy in Stroke Patients at High Risk of Developing Unprovoked Seizures: Anti-epileptogenic Effects of Eslicarbazepine Acetate
Brief Title: Anti-epileptogenic Effects of Eslicarbazepine Acetate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-213; 2018-002747-29 (EudraCT Number)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Post Stroke Epilepsy
Keywords: Prophylaxis; Post-stroke; Epilepsy; BIA 2-093; Unprovoked seizures; Eslicarbazepine acetate; Anti-epileptogenic; Bial - Portela & Ca, S.A.
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): ESL 800 mg
  Interventions: Drug: ESL 800 mg
- Group B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESL 800 mg — 800 mg ESL tablets for oral administration. In case a patient is unable to swallow the whole tablet, the tablet can be crushed or divided into equal doses at the score line.
  Other Names: Eslicarbazepine acetate, BIA 2-093
  Arms: Group A
Drug: Placebo — Placebo tablets for oral administration, matching the test product. In case a patient is unable to swallow the whole tablet, the tablet can be crushed or divided into equal doses at the score line.
  Arms: Group B

SUMMARY:
This study aims to assess if eslicarbazepine acetate (ESL) treatment (started within 96 hours after stroke occurrence and continued for 30 days) changes the incidence of unprovoked seizures (USs) within the first 6 months after randomisation as compared to placebo

DETAILED DESCRIPTION:
This is a multicentre, double-blind, randomised, placebo-controlled, parallel-group trial in patients with acute intracerebral haemorrhage with a Cortical involvement, Age <65 years, Volume of intracerebral haemorrhage > 10 ml and Early seizure within 7 days after intracerebral haemorrhage (CAVE) score ≥ 3 or an acute ischaemic stroke with a SeLECT score ≥ 6.

At the first visit (screening/baseline, V1a), patients will undergo several examinations to check eligibility. The next visit (V1b) has to be performed within 96 hours after primary stroke occurrence. After eligibility has been confirmed, patients will be randomised (randomisation ratio 1:1) to treatment with ESL 800 mg (Group A) or placebo (Group B).

Patients will start treatment with the investigational medicinal product (IMP), i.e. ESL or placebo, within 96 hours after primary stroke occurrence at V1b. They will continue treatment until Day 30 after randomisation and then be tapered off. Thereafter, patients will be followed up until 18 months after randomisation. Patients can concomitantly receive antiepileptic therapies, except commercially available ESL or oxcarbazepine, until Day 30.

Concomitant antiepileptic therapies have to be discontinued and down-titration has to be started according to the respective Summary of Product Characteristics (SmPC). If the antiepileptic drugs (AEDs)/benzodiazepine are not already discontinued before, downtitration must be started on Day 31 at the latest.

If one or more AS(s) occur(s) within 7 days after primary stroke, this will not result in change of IMP dose. Patients having a first US will discontinue IMP treatment and will be treated at the discretion of the investigator until 18 months after randomisation, except with commercially available ESL.

Further visits will be performed 7 days (V2, on-site), 37 days (V3, on-site), 12 weeks (V4, telephone), 26 weeks (V5, on-site), 38 weeks (V6, telephone), 52 weeks (V7, on-site), 64 weeks (V8, telephone) and 78 weeks (End of Trial (EoT) visit, on-site) after V1b.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

1. Male or female patient aged 18 years or above;
2. Acute intracerebral haemorrhage with a CAVE score ≥ 3 or acute ischaemic stroke with a SeLECT score ≥ 6, in each case confirmed by magnetic resonance imaging (MRI)/computed tomography (CT).
3. Time of stroke occurrence is known and V1b is planned within 96 hours.
4. Brain scan analysis has reliably excluded structural brain lesions that can mimic stroke, e.g. cerebral tumour or brain abscess, etc.
5. a. Patient is able to give informed consent and to write and has signed written informed consent OR b. Patient is able to give informed consent, but unable to write and has provided verbal witnessed consent OR c. Patient is unable to give informed consent, but likely to regain this ability until V2, and the informed consent is deferred OR d. Patient is unable to give informed consent, but likely to regain this ability until V2, and patient's legal representative (according to the respective national/local requirements) has provided written informed consent.
6. Female patients without childbearing potential (2 years postmenopausal, bilateral oophorectomy or tubal ligation, or complete hysterectomy) are eligible. Female patients with childbearing potential must not be pregnant as confirmed by a negative pregnancy test and sexually active females must use a medically acceptable effective nonhormonal method of contraception up to the end of the current menstrual cycle after stopping treatment. Acceptable methods for women are surgical intervention (e.g. bilateral tubal occlusion), intrauterine device, double-barrier methods, true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient) and vasectomised male partner, provided that he is the sole partner of that patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   Inclusion criteria at V1b
7. V1b is within 96 hours after stroke occurrence. Inclusion criteria at V2 (only applicable for patients who were unable to give informed consent at V1a.)
8. a. Patient is able to give informed consent and to write and has signed a written informed consent OR b. Patient is able to give informed consent, but unable to write and has provided verbal witnessed consent.

Exclusion Criteria:

Patients are to be excluded from the trial for ANY ONE of the following reasons:

1. Contraindication to ESL, i.e. known hypersensitivity to ingredients of ESL formulation or other carboxamide derivatives (e.g., oxcarbazepine, carbamazepine), or second or third degree atrioventricular (AV) block not corrected with a permanent pacemaker.
2. Known Han Chinese or Thai ancestry.
3. History of previous stroke (other than the one described in inclusion criteria no. 2 - 3).
4. Sinus venous thrombosis.
5. Spontaneous sub-arachnoid haemorrhage due to e.g. aneurysmatic or arteriovenous malformation.
6. History of USs prior to primary stroke.
7. Impaired pre-stroke level of function, i.e. modified Rankin Scale (mRS) score > 3 prior to first stroke occurrence.
8. History of AED use before primary stroke within the last 5 years as defined in the list of not allowed AEDs.
9. Use of ESL, unless provided as IMP of this trial, and oxcarbazepine.
10. Severe hepatic impairment.
11. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (measured at V1a).
12. Known or suspected acute or chronic alcoholism, delirium tremens, or toxic psychosis.
13. History of suicidal ideation or suicide attempt within the past 3 years.
14. Presence of any other significant or progressive/unstable medical condition that, in the opinion of the investigator, would compromise evaluation of the trial treatment or may jeopardise the patient's safety, compliance or adherence to protocol requirements, such as significant psychiatric, cardiovascular, respiratory, metabolic, endocrine, haematologic, infectious or neurological disease.
15. For women: Pregnancy or breast-feeding.
16. Previous enrolment in this trial or participation in any other investigational drug trial within the past 30 days (or 5 half-lives of IMP whichever is longer) prior to V1a.
17. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.
18. Employees of the investigator or trial centre, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial centre, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Trinka, MD MSc FRCP, Principal Investigator — Universitätsklinik für Neurologie; Matthias Koepp, MD PhD FRCP, Principal Investigator — UCL Institute of Neurology
Locations (22):
- Austria (5):
  - Klinikum am Wörthersee, Abteilung fur Neurologie, Klagenfurt, FeschnigstraBe 11
  - Medizinische Universität Innsbruck, Universitätsklinik für Neurologie, Innsbruck, Innrain 52
  - Kepler University Hospital, Med Campus III, Department of Neurology 2, Linz, Krankenhausstraße 9
  - Clinical Research Center Salzburg GmbH, Salzburg, Strubergasse 21
  - Kepler University Hospital GmbH, Neuromed Campus, Department of Neurology 1, Linz, Wagner-Jauregg-Weg 15
- Hospices Civils de Lyon, Neurological Hospitals, Bron, Boulevard Pinel, 59, France
- Germany (6):
  - UKGM Universitatsklinikum Marburg, Klinik und Poliklinik fur Neurologie, Marburg, Baldingerstrabe
  - Neurologische Universitatsklinik, Tübingen, Hoppe-Seyler-Strabe 3
  - Universitatsklinikum Essen, Klinik fur Neurologie, Essen, Hufelandstr. 55
  - LMU Ludwig-Maximilians-Universitat, Munchen, Klinikum Grobhadern, Neurologische Klinik und Poliklinik, Experimentelle Neurologie, München, Marchioninistrabe 15
  - Uniklinik RWTH Aachen, Klinik für Neurologie, Aachen, Pauwelsstr. 30
  - Universitatsklinikum Erlangen, Neurologische Klinik, Erlangen, Schwabachanlage 6
- Israel (2):
  - Sheba Medical Center, Neurology Department, Stroke Unit, Ramat Gan, Emek Ha'ella 1
  - Tel Aviv Sourasky Medical Center, Neurology Division, Tel Aviv, Weizmann 6
- Italy (3):
  - Clinica Neurologica e di Neuroriabllltazione - Azienda / Ospedallero-Universitarla S. Maria della Miserrcordia, Udine, P. Le S. Maria Della Misericordia, 15
  - Azienda Sanitaria Universitaria Integrata di Trieste - Ospedale Cattinara - Clinica Neurologica, Trieste, Strada Di Fiume 447
  - Azienda Sanitaria dell'Alto Adige - Ospedale di Merano, Merano, Via Rossini 5
- Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital Santa Maria - Serviço de Neurologia, Lisbon, Avenida Prof. Egas Moniz, Portugal
- Hospital Universitario Fundación Jiménez Diaz, Madrid, Avda. de Los Reyes Catolicos, 2, Spain
- Sahlgrenska universitetssjukhuset, Neurosjukvarden, Gothenburg, Bia Straket 7, Sweden
- United Kingdom (2):
  - King's College Hospital, London, Denmark Hill
  - Institute of Neurology, London, Queen Square

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4 patients failed screening. Overall, of 125 patients in the randomised set, 92 patients completed the 6-month period, 86 patients completed the 12-month period, and 84 patients completed the 18-month period. A total of 41 patients prematurely terminated the trial with similar frequencies in both treatment groups. Most of them terminated the trial before Visit 3 (24 patients) with lower frequency in the ESL group (10 patients) than in the placebo group (14 patients).
Period: Overall Study
Arm/Group | Group A | Group B
Started | 62 | 63
Safety Set | 61 | 62
Full Analysis Set | 61 | 62
Electroencephalogram (EEG) Analysis Subset | 31 | 34
Completed | 43 | 41
Not Completed | 19 | 22
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Consent was not given by the patient until V2 | 0 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 3 | 2
Not completed — Death | 4 | 0
Not completed — Stroke more than 7 days after primary stroke | 2 | 6
Not completed — Lost to Follow-up | 4 | 2
Not completed — Other. Not specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 27 | 57
  Between 18 and 65 years | 25 | 33 | 58
  >=65 years | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 38 | 40 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 57 | 60 | 117
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Female of childbearing potential [Count of Participants; unit: Participants] — Population: The percentage for females of childbearing potential is based on number of females
  Participants
    Yes: number analyzed (Participants) | 23 | 22 | 45
    Yes | 5 | 3 | 8
    No: number analyzed (Participants) | 23 | 22 | 45
    No | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experience the First Unprovoked Seizures (US) Within the First 6 Months After Randomisation (Failure Rate)
Description: Deaths before the first US or patients without evaluable assessment of the primary endpoint will be counted as treatment failures. To show that ESL (Group A) is superior to placebo (Group B), the primary null hypothesis will be tested against the alternative hypothesis
Time Frame: First 6 months after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Failures - Unprovoked seizure | 2 | 7
  Failures - Death | 3 | 0
  Failures - Withdrawn | 12 | 16
  Non-failures | 44 | 39

2. Secondary Outcome: Proportion of Patients Who Experience the First US During the First 12 Months After Randomisation
Description: as for outcome 1
Time Frame: First 12 months after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Failures - Unprovoked seizure | 3 | 8
  Failures - Death | 3 | 0
  Failures - Withdrawn | 13 | 18
  Non-failures | 42 | 36

3. Secondary Outcome: Proportion of Patients Who Experience the First US During the Course of the Trial
Description: as for outcome 1
Time Frame: Until 18 months after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Failures - Unprovoked seizure | 5 | 9
  Failures - Death | 4 | 0
  Failures - Withdrawn | 14 | 18
  Non-failures | 38 | 35

4. Secondary Outcome: Number of Acute Symptomatic Seizure (ASS)
Description: Number of ASSs will be summarised by means of descriptive statistics
Time Frame: During the first 7 days after stroke
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Patients without an ASS | 51 | 47
  Patients with at least one ASS | 10 | 15

5. Secondary Outcome: Probability of Failure at 6, 12, and 18 Months After Randomization
Description: The time to first US after randomisation will be analysed and presented by means of the Kaplan-Meier estimate after 6, 12 and 18 months for the failure time. The time to first US will be analysed from the day of randomisation.
Time Frame: Over 18 months follow-up period
Population: The time is related to 6, 12 and 18 months and the percentage means the estimated probability to experience a first US in that specific time.
Measure: Number; unit: Percentage of failure
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Percentage of failure
  Kaplan - Meier failure probability estimate at Month 6 (Day 182) | 3.50 | 14.55
  Kaplan - Meier failure probability estimate at Month 12 (Day 365) | 5.74 | 16.86
  Kaplan - Meier failure probability estimate at Month 18 (Day 547) | 10.34 | 19.17
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Other; p = 0.2081, Log Rank; Percentiles of time to first US = 92, 95% CI 2-sided [25 to 95]

6. Secondary Outcome: Time to First US After Stroke Occurrence.
Description: Analysis of time to first US will be performed using the day of stroke (before randomisation) as Day 1.
  The secondary objective and endpoint "Time to first US after stroke occurrence" was decided to be deleted as it is closely related to the forth secondary endpoint "Time to first US after randomisation" and therefore would not really have any additional value.
Time Frame: Over 18 months follow-up period
Population: Omitted with statistical analysis plan (SAP), Final version 1.0, 22-11-2023. Secondary objective and endpoint "Time to first US after stroke occurrence" was decided to be deleted as it is closely related to the forth secondary endpoint "Time to first US after randomisation" and therefore would not really have any additional value.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number and 4-week Rate of USs (4-week Rate of USs Was Omitted With SAP, Final Version 1.0, 22 NOV 2023).
Description: The total number and rate of USs, standardised per 4 weeks, in all patients and in patients with US(s) only will be summarised by means of descriptive statistics.
  The secondary objective and endpoint "4-week rate of USs" was decided to be deleted as this information will not be meaningful for this trial.
Time Frame: Over 18 months follow-up period
Population: Omitted with statistical analysis plan [SAP], Final version 1.0, 22-NOV-2023. Secondary objective and endpoint "Time to first US after stroke occurrence" was decided to be deleted as it is closely related to the forth secondary endpoint "Time to first US after randomisation" and therefore would not really have any additional value.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Barthel Index (BI) Original 10-item Version
Description: The Barthel Index at baseline and post-baseline visits of each patient will be calculated adding the individual scores from each item. Baseline is the value assessed before first IMP intake. Endpoint is the last non-missing value collected after the first IMP intake. The BI is a widely used score to measure the performance in activities of daily living of patients with stroke and other neuromuscular or musculoskeletal disorders in the following 10 categories:
  1. Feeding (scored as 0, 5, 10)
  2. Moving from a wheelchair to a bed and back again (scored as 0, 5, 10, 15)
  3. Personal hygiene (scored as 0, 5)
  4. Getting on and off the toilet (scored as 0, 5, 10)
  5. Self-bathing (scored as 0, 5)
  6. Walking on a level surface (scored as 0, 5, 10, 15)
  7. Ascending and descending stairs (scored as 0, 5, 10)
  8. Dressing (scored as 0, 5, 10)
  9. Controlling bowels (scored as 0, 5, 10)
  10. Controlling bladder (scored as 0, 5, 10) The minimum value means with help and maximum independent
Time Frame: Barthel Index data is collected at Baseline, V3 (+37 days), V5 (+26 weeks), V7 (+52 weeks), End of trial visit (EOT, +78 weeks) or Early discontinuation visit (EDV, on average 30 days), and Endpoint (18 months).
Population: The total BI score (possible range 0 - 100) will be calculated as the sum of the individual scores from each item.
  General ranges of BI describe patients' disability as follows:
  80-100 - patient should be able to live independently 60-79 - minimally dependent 40-59 - partially dependent 20-39 - very dependent <20 - total dependence
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Score on a scale
  Baseline - Observed Value | 66.1 [0 to 100] | 61.9 [0 to 100]
  V3 - Observed Value | 85.5 [0 to 100] | 87.2 [0 to 100]
  V5 - Observed Value | 94.3 [0 to 100] | 95.7 [0 to 100]
  V7 - Observed Value | 92.2 [0 to 100] | 96.3 [0 to 100]
  EDV - Observed Value | 66.0 [0 to 100] | 96.3 [0 to 100]
  EoT - Observed Value | 92.4 [0 to 100] | 94.9 [0 to 100]
  Endpoint | 87.5 [0 to 100] | 93.6 [0 to 100]

9. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficits.
  The following questions will be asked:
  1a. Level of Consciousness (LOC) (scored as 0, 1, 2, 3)
  1b. LOC Questions (scored as 0, 1, 2)
  1c. LOC Commands (scored as 0, 1, 2) 2. Best Gaze (scored as 0, 1, 2) 3. Visual (scored as 0, 1, 2, 3) 4. Facial Palsy (scored as 0, 1, 2, 3) 5a. Motor Arm (Left Arm) (scored as 0, 1, 2, 3, 4) 5b. Motor Arm (Right Arm) (scored as 0, 1, 2, 3, 4) 6a. Motor Leg (Left Leg) (scored as 0, 1, 2, 3, 4) 6b. Motor Right (Right Leg) (scored as 0, 1, 2, 3, 4) 7. Limb Ataxia (scored as 0, 1, 2) 8. Sensory (scored as 0, 1, 2) 9. Best Language (scored as 0, 1, 2, 3) 10. Dysarthria (scored as 0, 1, 2) 11. Extinction and Inattention (formerly Neglect) (scored as 0, 1, 2) The sum of all 15 individual scores will provide the patient's total NIHSS score where 0 is "no stroke symptoms" and 42 is "severe stroke".
Time Frame: National Institutes of Health Stroke Scale (NIHSS) data is collected at Baseline, V3 (+37 days), V5 (+26 weeks), V7 (+52 weeks), End of trial visit (EOT, +78 weeks) or Early discontinuation visit (EDV, on average 30 days), and Endpoint (18 months).
Population: Stroke severity will be stratified based on NIHSS total score as follows:
  <11 - mild and moderately severe
  ≥11 - severe
  For each patient, the total NIHSS score at baseline and each post-baseline visit will be calculated adding the individual scores from each item.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Score on a scale
  Baseline - Observed Value | 8.5 [0 to 42] | 8.8 [0 to 42]
  V2 - Observed Value | 4.6 [0 to 42] | 3.0 [0 to 42]
  V3 - Observed Value | 2.5 [0 to 42] | 1.5 [0 to 42]
  V5 - Observed Value | 1.9 [0 to 42] | 0.6 [0 to 42]
  V7 - Observed Value | 1.6 [0 to 42] | 0.8 [0 to 42]
  Early discontinuation visit - Observed Value | 3.4 [0 to 42] | 0 [0 to 42]
  End of trial visit - Observed Value | 1.5 [0 to 42] | 0.6 [0 to 42]
  Endpoint - Observed Value | 2.9 [0 to 42] | 1.5 [0 to 42]

10. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 can be used for screening, diagnosing and measuring the severity of depression in stroke patients. The patient will rate on a scale from 0 (not at all) to 3 (nearly every day) how often each of the 9 symptoms occurred during the past 2 weeks. The individual scores from each item of the PHQ-9 will be added to calculate the total PHQ-9 score for each time of examination.
Time Frame: Over 18 months follow-up period
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Points
  Baseline - Observed Value | 3.7 (3.34) | 3.4 (4.43)
  Endpoint - Observed Value | 4.1 (3.96) | 4.3 (5.25)
  Endpoint - Change from Baseline | 0.5 (4.61) | 0.7 (6.13)

11. Secondary Outcome: Overall Survival at 6, 12, and 18 Months After Randomization
Description: Overall survival (time to death relative to the date of randomization) will be analysed and presented by means of the Kaplan-Meier estimates (including censored data e.g. withdrawals) after 6 months (Day 182), 12 months (Day 365) and 18 months (Day 547) for the survival rates.
Time Frame: Over 18 months follow-up period
Population: Patients censored are all patients who discontinued the study due to any reason including death before study day 548.
  The time is related to 6, 12 and 18 months and the percentage means the probability to experience a first US in that specific time.
Measure: Number; unit: Percentage of death probability
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Percentage of death probability
  Kaplan - Meier death probability estimate at Month 6 (Day 182) | 5.64 | 0.00
  Kaplan - Meier death probability estimate at Month 12 (Day 365) | 5.64 | 0.00
  Kaplan - Meier death probability estimate at Month 18 (Day 547) | 7.74 | 0.00
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Other; p = 0.0542, Log Rank; Overall Survival

12. Secondary Outcome: Treatment Emergent Adverse Events (TEAEs) Incl. Findings From Physical and Neurological Examinations
Description: Adverse events (AEs) not considered treatment-emergent according to this definition or with missing data will be medically reviewed during the data review meeting and will be considered treatment emergent if appropriate
Time Frame: Over 18 months follow-up period
Population: TEAE: Adverse Event with onset or worsening after first IMP intake until 14 days after last IMP intake.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  TEAE | 50 | 51
  Non-serious TEAE | 50 | 48
  Serious TEAE | 12 | 13
  Related TEAE | 23 | 12
  Serious related TEAE | 3 | 0
  Severe TEAE | 9 | 8
  TEAE leading to discontinuation of IMP | 16 | 6
  TEAE leading to dose reduction | 0 | 2
  TEAE requiring medication | 36 | 46
  TEAE leading to death | 2 | 0
  Ongoing TEAE at the end of the trial | 31 | 30
  TEAE leading to study discontinuation | 4 | 4

13. Secondary Outcome: Clinically Significant Haematology Abnormalities
Description: Based on haemoglobin, haematocrit, red blood cell count (RBC), white blood cell count (WBC), differential - neutrophils, eosinophils, lymphocytes, monocytes and basophils, and platelet count. All laboratory values will be classified as normal or abnormal according to the laboratories normal ranges and as clinically significant according to the assessment of the investigator. For these tests, approximately 12 mL of blood will be collected at each blood withdrawal.
Time Frame: Over 18 months follow-up period
Population: Shifts of Haematology Parameters from Normal or Abnormal to Clinically Significant (CS) Abnormal at Endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Eosinophils - Low to CS high | 1 | 0
  Eosinophils abs. - Low to CS high | 1 | 0
  Lymphocytes - Low to CS low | 1 | 0
  Lymphocytes abs - Low to CS low | 1 | 0

14. Secondary Outcome: Clinically Significant Biochemistry Abnormalities, Including eGFR (Estimated Glomerular Filtration Rate) and Coagulation
Description: The biochemistry analysis is based on sodium (will be monitored for signs of hyponatraemia), potassium, chloride, calcium, phosphate, blood urea nitrogen, aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), alkaline phosphatase, creatine phosphokinase (CPK), creatinine, glucose, C-reactive protein, albumin, total protein, total cholesterol, low-density lipoproteincholesterol, high-density lipoprotein-cholesterol, triglycerides, and total bilirubin (bilirubin will be fractionated direct/indirect if elevated). eGFR will be estimated based on serum creatinine value using the according CKD-EPI formula using age, sex and race. Coagulation is based on international normalised ratio and activated partial thromboplastin time (aPTT). All laboratory values will be classified as normal or abnormal according to the laboratories normal ranges and as clinically significant according to the assessment of the investigator.
Time Frame: Over 18 months follow-up period
Population: Shifts of Biochemistry Parameters from Normal or Abnormal to Clinically Significant Abnormal at Endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Sodium - Normal to CS low | 1 | 0
  Potassium - Normal to CS low | 1 | 0
  Potassium - Normal to CS high | 1 | 0
  Potassium - Missing to CS high | 1 | 0
  Blood urea nitrogen - Missing to CS high | 1 | 0
  Aspartate transaminase - Normal to CS high | 1 | 0
  Alanine transaminase - Normal to CS high | 1 | 0
  Alanine transaminase - High to CS high | 1 | 0
  Gamma-glutamyl transferase - Normal to CS high | 3 | 0
  Lactate dehydrogenase - Low to CS high | 1 | 0
  Alkaline phosphatase - Normal to CS high | 2 | 1
  Creatinine - Normal to CS high | 1 | 1
  Creatinine - Missing to CS high | 1 | 0
  C-reactive protein - High to CS high | 2 | 0
  LDL-cholesterol - Normal to CS high | 1 | 0
  HDL-cholesterol - Normal to CS low | 2 | 0
  Triglycerides - Normal to CS high | 0 | 1
  Total bilirubin - Normal to CS high | 1 | 0
  Bilirubin direct - Missing to CS high | 1 | 0
  Glomerular filtration rate - Normal to CS low | 1 | 0
  International normalised ratio - High to CS high | 1 | 0
  Activated partial thromboplastin time - Normal to CS high | 2 | 0

15. Secondary Outcome: Clinically Significant Urinalysis Abnormalities
Description: The urinalysis is based on pH, specific gravity, protein, blood, glucose, ketones, bilirubin, urobilinogen (local dipstick). Microscopy and other appropriate tests (as needed) will be performed if dipstick indicates any significant abnormality. All laboratory values will be classified as normal or abnormal according to the laboratories normal ranges and as clinically significant according to the assessment of the investigator.
Time Frame: Over 18 months follow-up period
Population: The number analyzed are patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Clinically Significant abnormality - Baseline - No: number analyzed (Participants) | 60 | 56
  Clinically Significant abnormality - Baseline - No | 46 | 42
  Clinically Significant abnormality - Baseline - Yes: number analyzed (Participants) | 60 | 56
  Clinically Significant abnormality - Baseline - Yes | 14 | 14
  Clinically Significant abnormality - Endpoint - No: number analyzed (Participants) | 49 | 43
  Clinically Significant abnormality - Endpoint - No | 36 | 34
  Clinically Significant abnormality - Endpoint - Yes: number analyzed (Participants) | 49 | 43
  Clinically Significant abnormality - Endpoint - Yes | 13 | 9

16. Secondary Outcome: Clinically Significant Vital Sign Abnormalities: Blood Pressure
Description: The systolic and diastolic blood pressure (mmHg) were to be measured after the patient had rested for at least 5 minutes. Painful procedures, like drawing blood, had to be performed after vital signs measurements (not before). The analyses of variables for vital sign parameters will focus on the evaluation of the change from baseline to the scheduled time points after baseline. Descriptive statistics of the time course and of changes from baseline to each post-baseline time point will be presented by treatment group.
Time Frame: Over 18 months follow-up period
Population: Incidence of Clinically Significant Vital Sign Abnormalities at Baseline or Endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Systolic blood pressure [mmHg] - Baseline - CS high | 1 | 3
  Diastolic blood pressure [mmHg] - Baseline - CS low | 0 | 0
  Diastolic blood pressure [mmHg] - Baseline - CS high | 0 | 1
  Systolic blood pressure [mmHg] - Endpoint - CS high | 1 | 1
  Diastolic blood pressure [mmHg] - Endpoint - CS low | 0 | 1
  Diastolic blood pressure [mmHg] - Endpoint - CS high | 0 | 0

17. Secondary Outcome: Clinically Significant Vital Sign Abnormalities: Heart Rate
Description: The Heart Rate (bpm) were to be measured after the patient had rested for at least 5 minutes. Painful procedures, like drawing blood, had to be performed after vital signs measurements (not before). The analyses of variables for vital sign parameters will focus on the evaluation of the change from baseline to the scheduled time points after baseline. Descriptive statistics of the time course and of changes from baseline to each post-baseline time point will be presented by treatment group.
Time Frame: Over 18 months follow-up period
Population: Incidence of Clinically Significant Vital Sign Abnormalities at Baseline or Endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Pulse rate [bpm] - Baseline - CS high | 0 | 0
  Pulse rate [bpm] - Endpoint - CS high | 0 | 1

18. Secondary Outcome: Electrocardiogram (ECG)
Description: The ECG equipment is to be calibrated to 1 cm/mV and recording is to be done at 25 mm/sec and performed for a minimum of 10 sec. At V1a the investigator should examine the ECG for signs of cardiac disease that should exclude the patient from the trial. An assessment of normal or abnormal will be recorded and if the ECG abnormality is considered clinically significant, the abnormality will be documented in the electronic case report form (eCRF). If an ECG was done after primary stroke, the results should be used and the examination does not need to be repeated at V1a. After each recording of a simultaneous 12-lead resting ECG, a copy of the originally printed ECG records will be printed, assessed and filed by the investigator, in order to ensure that maintenance of the data will not be affected by thermolability of the paper.
Time Frame: A standard 12-lead electrocardiogram (ECG) is performed at Baseline, V2 (+7 days), V3 (+37 days), Early discontinuation visit (if EDV performed before V3, on average 30 days).
Population: The number analyzed are patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Participants
  Baseline - Clinically Significant abnormal: number analyzed (Participants) | 60 | 62
  Baseline - Clinically Significant abnormal | 9 | 8
  V2 - Clinically Significant abnormal: number analyzed (Participants) | 43 | 37
  V2 - Clinically Significant abnormal | 4 | 3
  V3 - Clinically Significant abnormal: number analyzed (Participants) | 34 | 32
  V3 - Clinically Significant abnormal | 4 | 3
  Early discontinuation visit - Clinically Significant abnormal: number analyzed (Participants) | 4 | 1
  Early discontinuation visit - Clinically Significant abnormal | 0 | 0
  Endpoint: number analyzed (Participants) | 47 | 41
  Endpoint | 4 | 3

19. Secondary Outcome: Suicidal Ideation and Behaviour, Assessed by PHQ-9 (Question 9)
Description: The individual scores from each item of the PHQ-9 will be added to calculate the total PHQ-9 score for each time of examination.Over the last 2 weeks, how often have you been bothered by any of the following problems?
  1. Little interest or pleasure in doing things
  2. Feeling down, depressed, or hopeless
  3. Trouble falling or staying asleep, or sleeping too much
  4. Feeling tired or having little energy
  5. Poor appetite or overeating
  6. Feeling bad about yourself - or that you are a failure or have let yourself or your family down
  7. Trouble concentrating on things, such as reading the newspaper or watching television
  8. Moving or speaking so slowly that other could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual
  9. Thoughts that you would be better off dead or of hurting yourself in some way The individual scores from each item of the PHQ-9 will be added to calculate the total PHQ-9 score for each time of examination.
Time Frame: The PHQ-9 will be collected at Baseline, V3 (+37 Days), V5 (+26 weeks), V7 (+52 weeks), End of trial visit (EOT, +78 weeks) or Early discontinuation visit (if EDV performed before V3, on average 30 days), and Endpoint (18 months).
Population: The patient will rate on a scale from 0 (not at all) to 3 (nearly every day) how often each of the 9 symptoms occurred during the past 2 weeks.
  The PHQ-9 total score will be categorised as follows:
  ≤4 - minimal depression >4 - mild to severe depression
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 61 | 62
Score on a scale
  Baseline - Observed Value: number analyzed (Participants) | 57 | 54
  Baseline - Observed Value | 3.7 (3.34) | 3.4 (4.43)
  V3 - Observed Value: number analyzed (Participants) | 49 | 44
  V3 - Observed Value | 5.0 (5.57) | 4.5 (5.12)
  V5 - Observed Value: number analyzed (Participants) | 41 | 43
  V5 - Observed Value | 5.0 (4.72) | 5.5 (5.91)
  V7 - Observed Value: number analyzed (Participants) | 39 | 36
  V7 - Observed Value | 3.9 (4.08) | 4.4 (5.12)
  Early discontinuation visit - Observed Value: number analyzed (Participants) | 4 | 4
  Early discontinuation visit - Observed Value | 2.0 (0.82) | 3.8 (4.35)
  End of trial visit - Observed Value: number analyzed (Participants) | 38 | 36
  End of trial visit - Observed Value | 3.8 (3.85) | 3.9 (5.50)
  Endpoint - Observed Value: number analyzed (Participants) | 53 | 48
  Endpoint - Observed Value | 4.1 (3.96) | 4.3 (5.25)

20. Secondary Outcome: Number of Participants With and Without Seizures Based on Electroencephalogram (EEG)
Description: Routine EEG assessment (standard 10-20 set of electrodes, digital recording with 256 Hz sampling rate) for a minimum of 20 min will be performed at the discretion of the investigator. The EEG will be performed as exploratory analysis to support the development of a predictor for the development of post-stroke epilepsy and is therefore an optional assessment. All EEG analyses will be presented for the EEG analysis subset (all patients in the full analysis set with a baseline and a post-baseline EEG recording available). EEG parameters will be evaluated exploratively using descriptive statistics.
  For this outcome was decided that results would be possibly explored in an manuscript.
Time Frame: Two recordings were provided: one carried out before in the initial phase of enrollment into the trial at V1a (< 96 hours) and the second one after termination of eslicarpazepine acetate intake (EOT, +78 weeks).
Population: The preprocessed EEG data was then analysed in two different ways; (i) we performed a power analyses and (ii) we calculated multivariate autoregressive models to investigate connectivity between channels. For both analyses the following frequency bands were defined and used to group the results: delta (1 - 3.9 Hz), theta (4 - 7.9 Hz), alpha (8 - 12.9 Hz), beta (13 - 39.9 Hz), gamma (>40Hz).
Measure: Count of Participants; unit: Participants
Groups:
- Group A: ESL 800 mg ESL 800 mg: 800 mg ESL tablets for oral administration. In case a patient is unable to swallow the whole tablet, the tablet can be crushed or divided into equal doses at the score line.
- Group B: Placebo Placebo: Placebo tablets for oral administration, matching the test product. In case a patient is unable to swallow the whole tablet, the tablet can be crushed or divided into equal doses at the score line.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 34
Participants
  EEG recordings of V1a - Patients with seizures | 16 | 24
  EEG recordings of EoT - Patients without seizures | 5 | 10
  Differences between EoT-V1a - Patients with seizures | 3 | 0
  Differences between EoT-V1a - Patients without seizures | 0 | 7

ADVERSE EVENTS:
Time Frame: The period of monitored/assessed for the collection of AEs started with the first onset or worsening after the first investigational medicinal product (IMP) intake at V1b until 14 days after the last IMP intake, up to 18 months per participant.
Description: Overall, 101 (82.1%) patients experienced TEAEs. Out of the 123 enrolled patients, 35 (28.5%) patients in total experienced at least one possibly related TEAE. Six deaths were reported. One patient died before randomisation and 5 patients who died were treated with ESL. One ESL group subject died but the primary reason for premature termination was "stroke more than 7 days after primary stroke" and not "intolerable AE" (including death).
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 6/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 12/61 | 13/62
Other Adverse Events (participants affected / at risk) | 50/61 | 48/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=61) | Group B (N=62)
Status epilepticus (Nervous system disorders) | 1 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral vasoconstriction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=61) | Group B (N=62)
Headache (Nervous system disorders) | 4 | 8
Dizziness (Nervous system disorders) | 4 | 0
Disturbance in attention (Nervous system disorders) | 2 | 1
Neuralgia (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral vasoconstriction (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 3 | 4
Anxiety (Psychiatric disorders) | 1 | 3
Agitation (Psychiatric disorders) | 1 | 2
Sleep disorder (Psychiatric disorders) | 2 | 1
Major depression (Psychiatric disorders) | 1 | 1
Post stroke depression (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 | 1
Sopor (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 13
Deep vein thrombosis (Vascular disorders) | 1 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 3
Hepatic enzyme increased (Investigations) | 2 | 1
High density lipoprotein decreased (Investigations) | 3 | 0
Blood creatinine increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Haemoglobin urine present (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Muscle enzyme increased (Investigations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 5
Candida infection (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Prostatic abscess (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 3 | 0
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 1
Feeling of body temperature change (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3
Cardiac failure (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT06597084/Prot_000.pdf
  • Statistical Analysis Plan: 0229_SAP_final_1.0_20231122 (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT06597084/SAP_001.pdf